CLINICAL TRIAL: NCT01890343
Title: A Study Evaluating the Imaging Characteristics of Florbetapir 18F (18F-AV-45) in Patients With Frontotemporal Dementia Compared to Patients With Alzheimer's Disease and Normal Controls.
Brief Title: Imaging Characteristics of Florbetapir 18F in Patients With Frontotemporal Dementia, Alzheimer's Disease and Normal Controls.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-010
Record Dates: First submitted 2013-06-27; First posted 2013-07-01 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer's Disease; Frontotemporal Dementia
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia | interventions — florbetapir; Fluorodeoxyglucose F18

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Frontotemporal Disorder (Experimental): Subjects with frontotemporal disorder (FTD) received a one-time intravenous (IV) bolus injection of 300 megabecquerels (MBq) florbetapir 18F and a one-time IV bolus injection of 185 MBq of 18F-FDG.
  Interventions: Drug: florbetapir 18F; Drug: 18F-FDG
- Cognitively Normal (Experimental): Cognitively normal (CN) subjects received a one-time intravenous (IV) bolus injection of 300 megabecquerels (MBq) florbetapir 18F.
  Interventions: Drug: florbetapir 18F
- Alzheimer's Disease (Experimental): Subjects with Alzheimer's disease (AD) received a one-time intravenous (IV) bolus injection of 300 megabecquerels (MBq) florbetapir 18F.
  Interventions: Drug: florbetapir 18F

INTERVENTIONS:
Drug: florbetapir 18F — Subjects received a one-time intravenous (IV) bolus injection of 300 megabecquerels (MBq) florbetapir 18F.
  Other Names: Florbetapir F 18; 18F-AV-45; Amyvid
Drug: 18F-FDG — FTD subjects received a one-time IV bolus injection of 185 MBq of 18F-FDG.
  Other Names: FDG; fluorodeoxyglucose (18F); fludeoxyglucose (18F)
  Arms: Frontotemporal Disorder

SUMMARY:
Study 18F-AV-45-010 is designed to evaluate the cerebral uptake of florbetapir 18F as measured by PET imaging in frontotemporal disorder (FTD) in comparison to cognitively normal volunteers and subjects with Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

AD:

* Male or female >= 50 years of age
* Meet National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) criteria for probable AD and have a Mini Mental State Examination (MMSE) score at screening between 10 and 24 inclusive
* Have a caregiver who can report on their mental status and activities of daily living (ADL)
* Give informed consent or have a caregiver give consent with subject assent.

FTD:

* Male or female >= 45 years of age
* Meet consensus criteria for FTD and have mild to moderate disease severity. Have a caregiver who can report on their mental status and ADL
* Give informed consent or have a caregiver give consent with subject assent.

CN:

* Male or female >= 45 years of age
* Have and MMSE >= 29
* Give informed consent

Exclusion Criteria:

* Have a history or a current clinically significant neurologic disease (other than AD or FTD, as applicable), a diagnosis of other dementing/neurodegenerative disease, or a diagnosis of mixed dementia
* Evidence from MRI or other biomarkers that suggests an etiology of dementia other than AD or FTD, as applicable or in the case of CN subjects evidence indicating the presence of AD, FTD or other types of neurologic pathology
* Have current clinically significant cardiovascular disease, screening ECG abnormalities, psychiatric disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, cancer or infectious disease
* Have a recent history of alcohol or substance abuse or dependence
* Women of childbearing potential who are not permanently surgically sterile, or are not refraining from sexual activity while not using adequate contraception.
* Require medications with a narrow therapeutic window, are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days
* Have ever participated in a study with an amyloid targeting agent
* Have had a radiopharmaceutical imaging or treatment procedure within 7 days of the imaging, other than as defined in the protocol

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (1):
- Research Site, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 subjects were enrolled in the trial but 6 subjects did not receive florbetapir and were not included in the Overall Study period.
Groups:
- Frontotemporal Disorder: Subjects with frontotemporal disorder (FTD).
  florbetapir 18F: Subjects received a one-time intravenous (IV) bolus injection of 300 megabecquerels (MBq) florbetapir 18F.
  18F-FDG: FTD subjects received a one-time IV bolus injection of 185 MBq of 18F-FDG.
- Cognitively Normal: Cognitively normal (CN) subjects.
  florbetapir 18F: Subjects received a one-time intravenous (IV) bolus injection of 300 megabecquerels (MBq) florbetapir 18F.
- Alzheimer's Disease: Subjects with Alzheimer's disease (AD).
  florbetapir 18F: Subjects received a one-time intravenous (IV) bolus injection of 300 megabecquerels (MBq) florbetapir 18F.
Period: Overall Study
Arm/Group | Frontotemporal Disorder | Cognitively Normal | Alzheimer's Disease
Started | 8 | 10 | 10
Completed | 8 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only subjects who received florbetapir (18F) are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Frontotemporal Disorder | Cognitively Normal | Alzheimer's Disease | Total
Number analyzed (Participants) | 8 | 10 | 10 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (9.62) | 62.4 (4.99) | 62.6 (4.35) | 62.5 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 3 | 8
  Male | 8 | 5 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 10 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Amyloid Image Assessment
Description: Four readers blinded to all clinical information classified florbetapir Positron Emission Tomography (PET) images as either positive for amyloid or negative for amyloid. The majority read classification is presented as either positive, negative or tied.
Time Frame: 50-60 min after injection
Measure: Number; unit: participants
Arm/Group | Frontotemporal Disorder | Cognitively Normal | Alzheimer's Disease
Number analyzed (Participants) | 8 | 10 | 10
participants
  Positive Scan | 2 | 1 | 8
  Negative Scan | 4 | 8 | 2
  Tie | 2 | 1 | 0

2. Primary Outcome: Quantitative Amyloid Image Assessment
Description: The effect of diagnostic group on mean total cortical grey matter florbetapir binding relative to cerebellar cortex is presented as standard uptake value ratios (SUVr).
Time Frame: 50-60 minutes after injection
Measure: Mean (Standard Deviation); unit: SUVr
Arm/Group | Frontotemporal Disorder | Cognitively Normal | Alzheimer's Disease
Number analyzed (Participants) | 8 | 10 | 10
SUVr | 1.25 (0.36) | 1.29 (0.11) | 1.77 (0.38)
Statistical Analysis 1: Comparison: Frontotemporal Disorder vs Cognitively Normal vs Alzheimer's Disease; The effect of diagnostic group on mean cortical florbetapir binding relative to cerebellar cortex was determined; Test type: Superiority or Other; p = 0.002, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Frontotemporal Disorder | Cognitively Normal | Alzheimer's Disease
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/8 | 0/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Frontotemporal Disorder (N=8) | Cognitively Normal (N=10) | Alzheimer's Disease (N=10)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days